CLINICAL TRIAL: NCT06507826
Title: Online Intervention Using Self-Compassionate Writing to Induce Positive Mood in Family Caregivers of Older Adults
Brief Title: Self-Compassionate Writing for Caregivers of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farah Wiita (Other)
Responsible Party: Sponsor-Investigator, Farah Wiita, PhD Candidate, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-193-AH
Record Dates: First submitted 2024-07-05; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Self-Compassion; Control
Keywords: Mindfulness; Self-kindness; Common humanity; Self-compassion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were unaware of condition assignment until after the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Control (Placebo Comparator): Descriptive writing.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Mindfulness (Active Comparator): Writing with mindfulness.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Mindfulness with Self-Kindness (Active Comparator): Writing with mindfulness and self-kindness.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Mindfulness with Common Humanity (Active Comparator): Writing with mindfulness and common humanity.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Control with Timed Response (Placebo Comparator): Descriptive writing.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Mindfulness with Timed Response (Active Comparator): Writing with mindfulness.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Self-Kindness with Timed Response (Active Comparator): Writing with self-kindness.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Common Humanity with Timed Response (Active Comparator): Writing with common humanity.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Revised Control (Placebo Comparator): Descriptive writing.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Self-Compassion (Active Comparator): Writing with mindfulness, self-kindness, and common humanity.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults
- Self-Compassion Without Mindfulness (Active Comparator): Writing with self-kindness and common humanity.
  Interventions: Behavioral: Self-Compassionate Writing for Caregivers of Older Adults

INTERVENTIONS:
Behavioral: Self-Compassionate Writing for Caregivers of Older Adults — Self-compassionate writing focusing on one or more self-compassion components (mindfulness, self-kindness, common humanity).

SUMMARY:
The goal of this study was to test an online writing intervention to encourage a self-compassionate mindset in family caregivers of older adults. The main aims were to answer the questions:

* Writing with self-compassion would increase self-compassion.
* Writing with self-compassion would improve mood. Researchers compared self-compassion components (self-kindness, which involves a gentle and non-judgemental approach to oneself at times of difficulty; common humanity, which includes recognising one's difficulties as part of a shared human experience; mindfulness, which includes noticing difficult feelings without becoming overwhelmed by them) to see which combinations achieved the best outcomes.

Participants wrote with different combinations of self-compassion components together, such as mindfulness and common humanity or mindfulness and self-kindness. Participants also wrote with self-kindness, common humanity, or mindfulness separately.

DETAILED DESCRIPTION:
After being informed and consenting to participate in the study, participants were allocated to a self-compassion or control condition. The study was designed to target state self-compassion and mood. The research was carried out over three studies, with refinements being made each time based on previous outcomes. In Studies 1 and 2, participants were tested for self-compassion and mood (guilt, sadness, and serenity). after the writing tasks. In Study 3, participants were asked to complete measures for these both before and after the writing tasks. The experiments were carried out online for all three studies.

ELIGIBILITY:
Inclusion Criteria:

* Family carer.
* Caring for a person over 65 years of age.
* Participants over 18 years of age.

Exclusion Criteria:

* Professional carers.
* Caring person under 65 years of age.
* Participants under 18 years of age.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Self-kindness measured with the State Self-Compassion Scale (Neff et al., 2021) | State measured immediately after intervention
  Scores closer to 5 expected on a scale of 1 to 5
Common humanity measured with the State Self-Compassion Scale (Neff et al., 2021) | State measured immediately after intervention
  Scores closer to 5 expected on a scale of 1 to 5
Mindfulness measured with the State Self-Compassion Scale (Neff et al., 2021) | State measured immediately after intervention
  Scores closer to 5 expected on a scale of 1 to 5

SECONDARY OUTCOMES:
Guilt measured using the Positive and Negative Affect Schedule (Watson and Clark, 1999) | State measured immediately after intervention
  Scores closer to 1 expected on a scale of 1 to 5
Sadness measured using the Positive and Negative Affect Schedule (Watson and Clark, 1999) | State measured immediately after intervention
  Scores closer to 1 expected on a scale of 1 to 5
Serenity measured using the Positive and Negative Affect Schedule (Watson and Clark, 1999) | State measured immediately after intervention
  Scores closer to 5 expected on a scale of 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Aileen K Ho, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data to be made available on OSF.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available on publication of the research report. It will be made available for 5 years.
Access Criteria: Access permitted under the conditions of the informed consent agreement.

REFERENCES:
- [Result] Neff, K. D., Tóth-Király, I., Knox, M. C., Kuchar, A., & Davidson, O. (2021). The development and validation of the state self-compassion scale (long-and short form). Mindfulness, 12, 121-140.
- [Result] Watson, David & Clark, Lee. (1999). The PANAS-X: Manual for the positive and negative affect schedule-expanded form. Psychology Publications.